CLINICAL TRIAL: NCT05035589
Title: The Effect of Tocilizumab on Procalcitonin and Other Biochemical and Clinical Markers in the Setting of COVID-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Sciberras, Stephen M.D. (Individual)
Collaborators: Mater Dei Hospital, Malta (Other)
Responsible Party: Principal Investigator, Stephen Sciberras, Investigator, Sciberras, Stephen M.D.
Other Study IDs: MDHITU-TCZ
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: COVID-19 Pneumonia; ARDS
Keywords: COVID-19 Pneumonia; Tocilizumab; Procalcitonin; C-Reactive Protein
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TCZ: The first 50 patients admitted to the ITU at Mater Dei Hospital with COVID-19 Pneumonia, to whom tocilizumab was administered
  Interventions: Drug: Tocilizumab
- Control: 50 patients admitted to ITU at Mater Dei Hospital with COVID-19 Pneumonia, who did not receive Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab administered at a dose of 8mg/kg up to a maximum of 800mg
  Groups: TCZ

SUMMARY:
This study aims to establish whether tocilizumab has any significant effect on procalcitonin levels on patients diagnosed with COVID-19 pneumonia requiring intensive care admission. The effects on other biochemical and clinical markers are also considered.

DETAILED DESCRIPTION:
A retrospective study, involving the first fifty patients treated with tocilizumab for acute deterioration in COVID-19 pneumonia in the Intensive Care Unit (ICU) at Mater Dei Hospital in Malta.

The following parameters will be collected from medical records:

* procalcitonin levels, daily for twenty days or until discharge or death.
* namely white cell count (WCC), neutrophils, lymphocytes,
* C-reactive protein (CRP)
* PaO2/FiO2 ratio (P/F ratio).

This group will be compared to a control group was chosen from patients admitted to the ICU who were not eligible for tocilizumab treatment, matched to the study group for age, gender, mode of ventilation required and length of stay in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 diagnosis
* Admitted to ITU
* Tocilizumab treatment

Exclusion Criteria:

* none

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 patients treated with tocilizumab single dose therapy in ICU
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Procalcitonin | throughout study completion, daily for maximum of 20 days
  effect of Tocilizumab on Procalcitonin levels

SECONDARY OUTCOMES:
CRP | throughout study completion, daily for maximum of 20 days
  effect of Tocilizumab on CRP levels
WCC | throughout study completion, daily for maximum of 20 days
  effect of Tocilizumab on WCC levels
Neutrophils | throughout study completion, daily for maximum of 20 days
  effect of Tocilizumab on Neutrophils levels
Lymphocytes | throughout study completion, daily for maximum of 20 days
  effect of Tocilizumab on Lymphocytes levels
NLR | throughout study completion, daily for maximum of 20 days
  effect of Tocilizumab on Neutrophil to Lymphocyte ratio
P/F ratio | throughout study completion, daily for maximum of 20 days
  effect of Tocilizumab on P/F ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Mater Dei Hospital, Msida, Malta

IPD SHARING:
Plan to Share IPD: Undecided